CLINICAL TRIAL: NCT06215378
Title: Antagonization of Heparin With Protamine Sulfate to Lower All Neurological Ischemic and Hemorrhagic Events After Transcatheter Aortic Valve Implantation for Aortic Stenosis
Brief Title: Antagonization of Heparin With Protamine Sulfate After TAVI
Acronym: ATLANTIS-Prota
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Action Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP211046
Record Dates: First submitted 2023-12-22; First posted 2024-01-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-01

CONDITIONS: Aortic Valve Stenosis; Heart Valve Diseases
Keywords: TAVI; Protamine; Heparine; Antagonization; Aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases | interventions — Protamines

STUDY DESIGN:
Intervention Model Description: Phase III, national, multicenter, controlled, randomized open label study in 2 parallel groups at a 1:1 ratio
Who Masked: Outcomes Assessor
Masking Description: The members of the endpoint committee will evaluate events related to both primary and secondary outcomes in a blinded manner, ensuring they are unaware of patient identities and the groups to which they were allocated through randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Systematic heparine antagonization with protamine sulphate (Experimental): Complete reversal of the Heparin administered during the TAVI achieved through the infusion of a protamine solution until the ACT returns to its baseline level.
  Interventions: Drug: Antagonization of heparin with protamine sulfate
- No Systematic heparine antagonization with protamine sulphate (No Intervention): No administration of protamine solution unless a participant encounters a bleeding event requiring a surgery or percutanous intervention.

INTERVENTIONS:
Drug: Antagonization of heparin with protamine sulfate — A systematic use at the end of procedure of Protamine Sulfate for antagonization of heparine.1 mg of protamine sulfate neutralizes approximately 100 heparin unit. To be administered in slow infusion (10 min) not exceeding 50mg of protamine sulfate to reverse 100% of the anti-IIa activity of heparin sodium. If the ACT is not back to the baseline value after the end of this infusion, additional doses of protamine should be performed depending on the ACT value to obtain complete antagonization of anti-IIa activity of heparin sodium
  Arms: Systematic heparine antagonization with protamine sulphate

SUMMARY:
Transcatheter aortic valve replacement (TAVR) is now the first therapeutic option offered to high and intermediate risk patients with symptomatic aortic stenosis but even to low-risk, when the aortic valve is tricuspid and the transfemoral approach is suitable. Vascular and bleeding complications are the most frequent procedure-related unwanted events associated with increased short-term morbidity and mortality. Selection of the appropriate vascular access site and pre-closing devices as well as stent implantation mitigate these complications.

ACT-guided heparin reaching a target of 300 seconds or more is recommended prior to the placement of the guiding sheath in the common femoral artery. Protamine sulfate is the heparin antidote, which antagonizes 100% of its anti-IIa activity and 60% of its anti-Xa activity. Reversal of heparin using protamine sulfate is recommended for transapical and complicated transfemoral aortic valve placement.However, there is a great heterogeneity of protamine use in daily practice and supportive evidence for the prevention of bleeding complications as well as its safety is lacking. In addition, the radial approach for the second vascular access is more commonly used as well as the use of echo-guided femoral puncture further questioning reversal of heparin when the procedure has been successfully completed without overt bleeding complications.

Our study aims to demonstrate the superiority of a strategy of systematic ACT-guided heparin administration followed by systematic antagonization with protamine sulfate over usual of care to reduce in-hospital mortality, vascular/bleeding complications, stroke and transcient ischemic attack, myocardial infarction or red blood cell transfusion, from randomization to hospital discharge

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age
* Any patient eligible for transfemoral TAVI, irrespective of the chronic antithrombotic treatment
* Written informed consent
* Registered at the French social healthcare

Exclusion Criteria:

* Any major protamine sulfate exposure contraindications defined as a history of severe pulmonary hypertension, acute pulmonary edema or history of bronchospasm related to protamine sulfate administration
* Known allergy to protamine sulfate
* Hypersensitivity to protamine sulfate including protamine contained as an excipient in NPH [Neutral Protamine Hagedorn] insulin, known protamine or protamine-heparine complex antibodies
* Non-femoral approach for the TAVI procedure
* Protamine sulfate exposure within 24h of randomization
* Fish allergy
* Mechanical valves
* For men: Sterile or Vasectomy
* Women of childbearing potential
* Pregnancy and breast feeding women
* Contemporaneous enrolment in an interventional clinical trial
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Composite of ischemic and bleeding events | From procedure to hospital discharge (or at 30 days whichever comes first)
  The primary endpoint is defined as the first occurrence, of any event of the composite of all-cause mortality, type 2, 3 or 4 bleeding, major or minor vascular complications, stroke or TIA, myocardial infarction or any redblood transfusion. The primary endpoint will be blindly determined by a clinical event committee according to the valve Academic Research Consortium-3 (VARC-3 classifications)

SECONDARY OUTCOMES:
In hospital stay | From procedure to hospital discharge, assessed up to 30 days
  Assessment of length of in-hospital stay in days post TAVI procedure
Bleeding complication | From procedure to hospital discharge (or at 30 days whichever comes first)
  Assessment of the occurrence of:
  * Type 2, 3 or 4 bleeding according to the VARC 3 criteria or any red blood cell transfusion of minor or vascular complications.
  * Type 2, 3 or 4 bleedings or red blood cell transfusion.
  * Any red blood cell transfusion
  * Type 2, 3 or 4 bleedings
Assessement of interaction | From procedure to hospital discharge (or at 30 days whichever comes first)
  Assessment of an interaction in the impact of systematic antagonization according to the use or not of an echo-guided femoral puncture and/or arterial radial access. These subgroups are defined at the time of randomization by stratification.
Assessement of adverse outcome | From procedure to hospital discharge (or at 30 days whichever comes first)
  Assessment of the occurrence of:
  * Death or type 2, 3 or 4 bleedings
  * Any kidney injury, stage 2 to 4 according to the KDIGO definition
  * Death, type 2, 3 or 4 bleedings or stroke
  * Death, VARC 3 type 2-3-4 bleeding or Any red blood cell transfusion, MI or stroke Or TIA
  * Any myocardial infarction, stroke or TIA
  * Type 3 or 4 bleeding
  * Type 2 bleeding
  * Minor vascular complications
  * Access site and access related vascular injury according to VARC-3 criteria
Assessement of long term adverse outcome | From procedure 12 months post procedure
  Assessment of the composite of: Death, stroke, TIA, MI and bleeding VARC type 2 or more as well as each individual endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié Salpêtrière hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided